CLINICAL TRIAL: NCT03785366
Title: A Randomized, Single-Blind, Comparative Bioavailability Study to Assess the Pharmacokinetic Properties of VeraCept® Intrauterine Contraceptive vs ParaGard® in Healthy, Post-Menarcheal Women
Brief Title: A PK Study Comparing VeraCept vs. ParaGard Intrauterine Devices (IUDs)
Acronym: IUD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sebela Women's Health Inc. (Industry)
Collaborators: Synteract, Inc. (Industry)
Responsible Party: Sponsor
Organization: Sebela Pharmaceuticals Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CMDOC-0045
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Women at Risk for Pregnancy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects are blinded until the Day 57 Visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VeraCept (Experimental): VeraCept subjects will be inserted with VeraCept on Day 1. At Day 57 subjects will be informed that they received VeraCept and may continue in the study for up to 5 years
  Interventions: Drug: VeraCept
- ParaGard (Active Comparator): ParaGard subjects will be inserted with ParaGard on Day 1. At Day 57 subjects will be informed that they received ParaGard and may choose to have the ParaGard removed or continue use per standard of clinical care.
  Interventions: Drug: ParaGard

INTERVENTIONS:
Drug: VeraCept — VeraCept Intrauterine Device (IUD)
  Arms: VeraCept
Drug: ParaGard — ParaGard intrauterine copper contraceptive
  Other Names: ParaGard T 380A
  Arms: ParaGard

SUMMARY:
to Assess the Pharmacokinetic Properties of VeraCept® Intrauterine Contraceptive vs ParaGard® in Healthy, Post- Menarcheal Women

ELIGIBILITY:
Inclusion Criteria:

* Post-menarcheal, pre-menopausal females up to 45 years of age at the time of informed consent/assent and in good general health;
* History of regular menstrual cycles defined as occurring every 21-35 days when not using hormones or prior to recent pregnancy or spontaneous or induced abortion;
* Sexually active with a male partner who has not had a vasectomy;
* Reasonably expect to have coitus at least once monthly during the study period;
* In a mutually monogamous relationship of at least 3 months duration;
* Seeking to avoid pregnancy for the duration of the study;
* Willing to use the study drug as the sole form of contraception;
* Willing to accept a risk of pregnancy;
* Subjects who are age 21 or older, at time of informed consent, must have a normal papanicolaou test (Pap) or atypical squamous cells of undetermined significance (ASC-US) with negative high risk human papilloma virus (HPV) test result within the appropriate screen timeframe per American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines, and prior to the study IUD insertion. Alternatively, the subject must have had a colposcopy performed within the appropriate screen timeframe, and prior to the study IUD insertion that showed no evidence of dysplasia requiring treatment per ASCCP guidelines, or treatment was performed and follow-up at least 6 months after the treatment showed no evidence of disease by clinical evaluation;
* Able and willing to comply with all study tests, procedures, assessment tools and follow-up;
* Able and willing to provide and document informed consent and Authorization for Release of Protected Health Information (PHI). Unemancipated subjects under 18 years old must provide assent and have written parental consent documented on the consent form consistent with local legal requirements;
* Plan to reside within a reasonable driving distance of a research site for the duration of the study.
* Subject agrees not to self-remove VeraCept

Exclusion Criteria:

* Known or suspected pregnancy; or at risk for pregnancy from unprotected intercourse earlier in current cycle;
* A previously inserted intrauterine device (IUD) that has not been removed by the time the study IUD is placed;
* History of previous IUD complications, such as perforation, expulsion, or pregnancy with IUD in place;
* Pain with current IUD;
* Use of ParaGard IUD within the past 3 months
* Planned use of any non-contraceptive estrogen, progesterone or testosterone any time during the 60 months of study participation;
* Exclusively breastfeeding before return of menses; lactating women will be excluded unless they have had 2 normal menstrual periods prior to enrollment;
* Unexplained abnormal uterine bleeding (suspicious for a serious condition), including bleeding 4 weeks post-septic abortion or puerperal sepsis;
* Severely heavy or painful menstrual bleeding;
* Suspected or known cervical, uterine or ovarian cancer, or unresolved clinically significant abnormal Pap smear requiring evaluation or treatment;
* Any history of gestational trophoblastic disease with or without detectable elevated ß-human chorionic gonadotropin (ß-hCG) levels, or related malignant disease;
* Any congenital or acquired uterine anomaly that may complicate study drug placement, such as:

  * Submucosal uterine leiomyoma
  * Asherman's syndromes
  * Pedunculated polyps
  * Bicornuate uterus
  * Didelphus or uterine septa
* Any distortions of the uterine cavity (e.g. fibroids), that, in the opinion of the investigator, are likely to cause issues during insertion, retention or removal of the IUD;
* Untreated acute cervicitis or vaginitis within the past 3 months;
* Known or suspected human immunodeficiency virus (HIV) infection or clinical AIDS;
* Subjects who have an established immunodeficiency;
* Known intolerance or allergy to any components of VeraCept or ParaGard including intolerance or allergy to nickel, titanium, or copper, and including Wilson's Disease;
* Currently participating or planning future participation in a research study of an investigational drug or device during the course of this investigational study. Subject must have waited at least 30 days from exiting their last study prior to informed consent in this study;
* Subject has been enrolled in a previous VeraCept study;
* Known or suspected alcohol or drug abuse within 12 months prior to the screening visit;
* Any general health, mental health or behavioral condition that, in the opinion of the investigator, could represent an increased risk for the subject or would render the subject less likely to provide the needed study information;
* Study staff or a member of the immediate family of study staff.
* Concurrent use of corticosteroids

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 41 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, MPH, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - OHSU Women's Health Research Unit, Portland, Oregon
  - Seattle Women's Health, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VeraCept | ParaGard
Started | 21 | 20
Successful IUD Insertion | 20 | 19
Early Terminations | 1 | 2
Completed | 19 | 17
Not Completed | 2 | 3
Not completed — Non-Menstrual Pelvic Pain | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Partial IUD Expulsion | 0 | 2
Not completed — Unsuccessful IUD Insertion | 0 | 1

BASELINE CHARACTERISTICS:
Population: Number of participants who had a successful IUD insertion
Groups:
- Total: Total of all reporting groups
Arm/Group | VeraCept | ParaGard | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (6.42) | 29.9 (6.57) | 28.4 (6.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 11 | 12 | 23
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (5.82) | 25.6 (6.70) | 25.9 (6.19)
Height [Mean (Standard Deviation); unit: cm] | 166 (8.65) | 167 (6.27) | 166 (7.49)
Weight [Mean (Standard Deviation); unit: kg] | 72.6 (18.2) | 71.4 (20.4) | 72.0 (19.1)

OUTCOME MEASURES:

1. Primary Outcome: Relative Maximum Observed Total Serum Copper Concentration of VeraCept vs ParaGard (Cmax)
Description: Assess the relative bioavailability of observed systemic copper from VeraCept versus ParaGard based on Cmax
Time Frame: Study Days Baseline (pre-insertion), 3, 8, 15, 22, 29, 57
Population: One subject in the ParaGard group discontinued from the study prior to collection of the first post-insertion sample. Therefore, the overall number of participants analyzed in the ParaGard group differs from the overall number of baseline participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VeraCept | ParaGard
Number analyzed (Participants) | 20 | 18
ng/mL | 1210 (202) | 1300 (217)
Statistical Analysis 1: Comparison: VeraCept vs ParaGard; Test type: Other — For the primary analysis, a ANOVA model with treatment as a fixed effect and subject as a random effect was used to analyze the uncorrected PK parameters Cmax, Cmean, and AUC0-56 days. Analysis methodology for the secondary analysis mirrored the approach for the primary analysis applied to the baseline-corrected PK parameters; ANCOVA; test to Reference geometric mean ratio = 0.930, 90% CI 2-sided [0.80 to 1.25]

2. Primary Outcome: Mean Serum Concentration of Copper for VeraCept vs. ParaGard (Cmean)
Description: Assess the relative bioavailability of observed systemic copper from VeraCept versus ParaGard based on Cmean
Time Frame: Study Days Baseline (pre-insertion), 3, 8, 15, 22, 29, 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VeraCept | ParaGard
Number analyzed (Participants) | 20 | 18
ng/mL | 1070 (155) | 1150 (151)

3. Primary Outcome: Maximum Serum Concentration of Copper for VeraCept vs. ParaGard (AUC0-56)
Description: Assess the maximum relative bioavailability of observed systemic serum levels of copper from VeraCept versus ParaGard based on AUC0-56
Time Frame: From Baseline (pre-insertion) through the last measurable non-zero concentration, up to Day 57 (56 days post-insertion), with a minimum of 50 days post-insertion required for inclusion.
Population: Four subjects (2 in VeraCept group, 2 in ParaGard group) did not meet the minimum number of days for inclusion in the analyses. Therefore, the overall number of participants analyzed in each group differs from the overall number of baseline participants
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | VeraCept | ParaGard
Number analyzed (Participants) | 18 | 17
day*ng/mL | 59700 (8310) | 63600 (8130)

4. Secondary Outcome: Baseline-corrected Maximum Total Serum Copper Concentration of VeraCept vs. ParaGard (Cmax)
Description: To assess the relative bioavailability of baseline-corrected maximum total serum copper concentration of from the VeraCept IUD versus ParaGard based on Cmax
Time Frame: Study Days Baseline (pre-insertion), 3, 8, 15, 22, 29, 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VeraCept | ParaGard
Number analyzed (Participants) | 20 | 18
ng/mL | 63.5 (84.1) | 83.2 (70.6)

5. Secondary Outcome: Baseline-corrected Mean Total Serum Copper Concentration of VeraCept vs. ParaGard (Cmean)
Description: To assess the relative bioavailability of baseline-corrected mean total serum copper concentration of VeraCept IUD versus ParaGard based on Cmean
Time Frame: Study Days Baseline (pre-insertion), 3, 8, 15, 22, 29, 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VeraCept | ParaGard
Number analyzed (Participants) | 20 | 18
ng/mL | 15.0 (21.2) | 27.7 (27.3)

6. Secondary Outcome: Baseline-Corrected Maximum Serum Concentration of Copper for VeraCept vs. ParaGard (AUC0-56)
Description: To assess the relative bioavailability of baseline-corrected total serum copper from the VeraCept IUD versus ParaGard based on AUC0-56 days
Time Frame: Study Days Baseline (pre-insertion), 3, 8, 15, 22, 29, 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day*ng/ml
Arm/Group | VeraCept | ParaGard
Number analyzed (Participants) | 20 | 18
day*ng/ml | 992 (1680) | 1620 (1700)

7. Secondary Outcome: Total Serum Copper Levels of VeraCept vs. ParaGard Compared to Normal Copper Levels
Description: To assess the total serum copper levels within each treatment relative to the normal range (49 to 184 µg/dL).
Time Frame: Study Days Baseline (pre-insertion), 3, 8, 15, 22, 29, 57 (VeraCept and ParaGard), Months 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 (VeraCept only)
Population: One subject in the ParaGard group discontinued from the study prior to collection of the first post-insertion sample and is not included in this table. Therefore, the overall number of participants analyzed in the ParaGard group differs from the overall number of baseline participants.
Measure: Count of Participants; unit: Participants
Arm/Group | VeraCept | ParaGard
Number analyzed (Participants) | 20 | 18
Participants
  Baseline: Low | 0 | 0
  Baseline: Normal | 20 | 18
  Baseline: High | 0 | 0
  Day 3: Low | 0 | 0
  Day 3: Normal | 20 | 17
  Day 3: High | 0 | 1
  Day 8: Low | 0 | 0
  Day 8: Normal | 20 | 18
  Day 8: High | 0 | 0
  Day 15: Low | 0 | 0
  Day 15: Normal | 20 | 18
  Day 15: High | 0 | 0
  Day 22: number analyzed (Participants) | 19 | 17
  Day 22: Low | 0 | 0
  Day 22: Normal | 19 | 17
  Day 22: High | 0 | 0
  Day 29: number analyzed (Participants) | 20 | 17
  Day 29: Low | 0 | 0
  Day 29: Normal | 20 | 17
  Day 29: High | 0 | 0
  Day 57: number analyzed (Participants) | 18 | 17
  Day 57: Low | 0 | 0
  Day 57: Normal | 18 | 17
  Day 57: High | 0 | 0
  Month 6: number analyzed (Participants) | 18 | 0
  Month 6: Low | 0 |
  Month 6: Normal | 18 |
  Month 6: High | 0 |
  Month 12: number analyzed (Participants) | 17 | 0
  Month 12: Low | 0 |
  Month 12: Normal | 17 |
  Month 12: High | 0 |
  Month 18: number analyzed (Participants) | 15 | 0
  Month 18: Low | 0 |
  Month 18: Normal | 15 |
  Month 18: High | 0 |
  Month 24: number analyzed (Participants) | 15 | 0
  Month 24: Low | 0 |
  Month 24: Normal | 15 |
  Month 24: High | 0 |
  Month 30: number analyzed (Participants) | 12 | 0
  Month 30: Low | 0 |
  Month 30: Normal | 12 |
  Month 30: High | 0 |
  Month 36: number analyzed (Participants) | 11 | 0
  Month 36: Low | 0 |
  Month 36: Normal | 11 |
  Month 36: High | 0 |
  Month 48: number analyzed (Participants) | 11 | 0
  Month 48: Low | 0 |
  Month 48: Normal | 11 |
  Month 48: High | 0 |
  Month 60: number analyzed (Participants) | 8 | 0
  Month 60: Low | 0 |
  Month 60: Normal | 8 |
  Month 60: High | 0 |

8. Secondary Outcome: Long-term Stability of Copper Levels as Determined by Cmax - VeraCept Only
Description: To assess the long-term stability of copper levels following insertion of the VeraCept IUD
Time Frame: Study Days Baseline (pre-insertion), 3, 8, 15, 22, 29, 57, Months 6, 12, 18, 24, 30, 36, 42, 48, 54, 60
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VeraCept
Number analyzed (Participants) | 20
ng/mL | 87.3 (92.4)

9. Secondary Outcome: Long-term Stability of Copper Levels as Determined by Cmean - VeraCept Only
Description: To assess the long-term stability of copper levels following insertion of the VeraCept IUD
Time Frame: Study Days Baseline (pre-insertion), 3, 8, 15, 22, 29, 57, Months 6, 12, 18, 24, 30, 36, 48, 60
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VeraCept
Number analyzed (Participants) | 20
ng/mL | 18.7 (24.9)

ADVERSE EVENTS:
Time Frame: 5 years (60 months) for VeraCept, D57 for ParaGard
Arm/Group | VeraCept | ParaGard
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 19/20 | 8/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VeraCept (N=20) | ParaGard (N=19)
Intermenstrual bleeding (Reproductive system and breast disorders) | 8 (12) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 5 (5) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 2 (3) | 1 (1)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervix inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Coital bleeding (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vulvovaginal rash (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 2 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Athetosis (Nervous system disorders) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 0 (0)
Device expulsion (Product Issues) | 0 (0) | 2 (2)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal odour (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (3) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Papilloma viral infection (Infections and infestations) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Smear cervix abnormal (Investigations) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT03785366/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03785366/SAP_001.pdf